CLINICAL TRIAL: NCT06536205
Title: The Effect of Acceptance Commitment Therapy Based Psychoeducation on Hope, Resilience and Stress Levels in Individuals Experiencing Earthquake
Brief Title: Acceptance-commitment Therapy-based Psychoeducation for Individuals Experiencing Earthquakes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Collaborators: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Hacer Kabakoğlu, Lecturer, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Hacer.. MustafaKU
Record Dates: First submitted 2024-07-31; First posted 2024-08-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Violent Traumatic Event Having Been in an Earthquake (History)
Keywords: earthquake; psychological resilience; hope; stress

STUDY DESIGN:
Intervention Model Description: There is an experimental and a control group in the research.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): An 8-week training based on acceptance and commitment therapy will be applied to this group.
  Interventions: Behavioral: psychoeducation
- control group (No Intervention): There will be no intervention in this group. Only relevant forms will be filled out.

INTERVENTIONS:
Behavioral: psychoeducation — Psychoeducation, psychological difficulties or physical diseases; These are structured educational interventions aimed at teaching people about their illness and their emotional responses to the illness, developing coping skills, ensuring compliance with the illness and cooperation with treatment.
  Arms: experimental group

SUMMARY:
This research aims to reduce the stress level of individuals within the scope of acceptance and determination-based psychoeducation, to increase the individual's positive expectations for the future, to increase the sense of hope, which represents the individual's belief in the world and his thoughts that life is worth living, and to increase the individual's adaptation and coping skills after negative situations. It is aimed to increase the defined psychological resilience. The research is planned to be carried out with individuals registered in Bursa-Kütahya container city and Qatar-2 Container city in Hatay Antakya District and who experienced the earthquake centered in Kahramanmaraş on February 6, 2023. The population of the research will consist of individuals who experienced the earthquake registered in Bursa Kütahya container city and Qatar-2 container city. The sample of the research will consist of 40 people living in Bursa Kütahya container city and Qatar-2 container city and agreeing to participate in the research. The experimental group will be composed of 60 people, while 40 people will constitute the control group. In both groups, an introductory information form, Dispositional Hope Scale, The Brief Resilience Scale and Posttraumatic Diagnostic Scale will be applied to individuals with face-to-face interview technique and the answers given by the individuals will be recorded. After 8 weeks of acceptance and commitment-based psychoeducation is given to the experimental group, the forms used in the research will be re-administered to both the experimental group and the control group. Follow-up will be done 3 months after the last session of the training. The research will be conducted as a randomized controlled experimental. The research is planned between March 2024 and 20 September 2024.

DETAILED DESCRIPTION:
Earthquake is a natural event that causes social consequences by causing physical, economic and social psychological losses in addition to environmental damage in the region where it occurs. The February 6 Kahramanmaraş earthquake that we experienced in our recent history has been described as the disaster of the century. 13.5 million people were affected by the earthquake and 50 thousand people died. In Hatay, one of the earthquake regions, 22 thousand people lost their lives and 6 thousand 369 buildings were destroyed. People lost their relatives and friends, and many people either lost their limbs or lost their physical integrity during the disaster. The fact that individuals had difficulty finding their relatives after the earthquake and that almost every individual lost someone from their family, friend or circle further deepened the trauma. Therefore, timely and appropriate psychosocial assistance is important for disaster victims. High quality standards and guidance for care providers, ideally using evidence-based procedures, are important. One of the psychosocial interventions to be used for trauma is psychoeducation. This psychoeducation for recovery from trauma involves helping a person understand how exposure to traumatic threat(s) may affect their functioning, how to reduce these effects, and ways to bounce back from these experiences. The two most important goals of psychoeducation are: (a) to increase understanding of common responses to trauma, (b) to help "normalize" these responses as understandable responses to abnormal situations. Other goals are to teach effective coping techniques and to identify more severe or prolonged reactions that may require more intensive help or treatment. In this research, psychoeducation based on Acceptance and Commitment Therapy, one of the new methods, will be used. Acceptance and commitment therapy is a member of the family of psychotherapy approaches defined as cognitive-behavioral therapies and recommends revealing the relationship between cognition and behavior with empirical data, without ignoring the importance of cognitions in achieving behavioral change. This research aims to reduce the stress level of individuals within the scope of acceptance and determination-based psychoeducation, to increase the individual's positive expectations for the future, to increase the sense of hope, which represents the individual's belief in the world and his thoughts that life is worth living, and to increase the individual's adaptation and coping skills after negative situations. It is aimed to increase the defined psychological resilience. The research is planned to be carried out with individuals registered in Bursa-Kütahya container city and Qatar-2 Container city in Hatay Antakya District and who experienced the earthquake centered in Kahramanmaraş on February 6, 2023. The population of the research will consist of individuals who experienced the earthquake registered in Bursa Kütahya container city and Qatar-2 container city. The sample of the research will consist of 60 people living in Bursa Kütahya container city and Qatar-2 container city and agreeing to participate in the research. The experimental group will be composed of 60 people, while 60 people will constitute the control group. In both groups, an introductory information form, Dispositional Hope Scale, The Brief Resilience Scale and Posttraumatic Diagnostic Scale will be applied to individuals with face-to-face interview technique and the answers given by the individuals will be recorded. After 8 weeks of acceptance and commitment-based psychoeducation is given to the experimental group, the forms used in the research will be re-administered to both the experimental group and the control group. Follow-up will be done 3 months after the last session of the training. The research will be conducted as a randomized controlled experimental. The research is planned between March 2024 and 20 September 2024.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age.
* Being literate.
* Agreeing to participate in the study
* Having experienced the February 06 Turkey-Syria centered earthquake.
* Living in Hatay-Antakya Bursa Kütahya Container City or Qatar-2 container city.
* There is no obstacle to communication.

Exclusion Criteria:

* Having any mental illness.
* Having any mental or intellectual disorder.
* Illiteracy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-08-21 (Estimated)

PRIMARY OUTCOMES:
Acceptance-commitment therapy-based psychoeducation | 2 months
  Individuals living in container cities and willing to participate in the study were identified. Experimental and control groups were determined among these individuals by randomization method. Training was given to the experimental group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided